CLINICAL TRIAL: NCT05991570
Title: Uni-portal Thoracoscopic Exploration in Comparison to Exploratory Thoracotomy in Hemodynamically Stable Thoracic Trauma Patients
Brief Title: Thoracoscopic Exploration in Comparison to Exploratory Thoracotomy in Chest Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Hussein Rushdi, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AssiutCTS
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Thoracic Injury
MeSH Terms: conditions — Thoracic Injuries | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Intervention Model Description: cohort study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Other): Use of vedio assisted thoracoscopic surgery in exploration in diagnosis and treatment of chest trauma patients whos heamodynamically stable
  Interventions: Procedure: Video Assisted Thoracoscopic Surgery (VATS)
- control (Other): exploratory thoracotomy inchest trauma patients in failure of vedio assisted thoracoscopic surgery or in haemodynamically instable patients
  Interventions: Procedure: Video Assisted Thoracoscopic Surgery (VATS)

INTERVENTIONS:
Procedure: Video Assisted Thoracoscopic Surgery (VATS) — VATS is minimally invasive procedure for exploration to diagnose and treat thoracic injuries alternative to exploratory thoracotomy.
  Other Names: Thoracoscopic Exploration

SUMMARY:
Video-assisted thoracic surgery has a standard role in diagnosis and therapy in thoracic surgery, In the past, most patients necessitating surgical treatment secondary to chest trauma was exposed to open thoracotomy, which was the most morbid of surgical incisions

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery has become a popular and acceptable method for diagnosis of intra-thoracic lesions since 1990s with the developments in surgical techniques. It is also used for treatment of retained pleural collections, it is a simple alternative to open thoracotomy. Although it's multiple advantages, timing of surgery and its effects on patients' results are not well elucidated. Multiple studies report that prognosis of patients is better with the earlier interventions in injured chest. However, there is so many differences for the optimal time for surgery in these studies .

Indications of VATS have been extended for management of diagnosis and treatment of chest trauma since 1990. This approach has multiple advantages as chest tube setting, minimally invasive surgery, less postoperative pain, and chest exploration. Today, VATS is used for empyema, persistent pneumothorax, retained haemothorax, mediastinal and diaphragmatic exploration, pleuro-pericardial ruptures, surgery for thoracic duct injury and aspiration of symptomatic foreign bodies.

ELIGIBILITY:
Inclusion Criteria:

1. patient aged more than 13 yards old
2. Hemo-dynamically stable patients with chest trauma
3. Willing and able to provide written informed consent and comply with study requirements.

Exclusion Criteria:

1. patient aged less than 13 yards old.
2. Hemo-dynamically instable patients
3. Head trauma patients.
4. missing informed consent
5. Participation in another clinical research.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Duration of airleak, lung expansion and post operative bleeding. | 2 weaks postoperative
  • Duration of complete healing: By
  1. Radiological (chest x-ray ant-post view and lat view & MSCT chest post-operative.
  2. Clinical examination post operative.

IPD SHARING:
Plan to Share IPD: No
through international publication